CLINICAL TRIAL: NCT07196150
Title: Comparison of the Effects of Exercise, Motor Imagery Training, and Pain Neuroscience Education on Pain, Menstrual Symptoms, and Cognitive Flexibility in Women With Primary Dysmenorrhea: A Randomized Controlled Trial
Brief Title: Exercise, Motor Imagery, and Pain Neuroscience Education for Primary Dysmenorrhea: A Randomized Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muge Dereli (Other)
Responsible Party: Sponsor-Investigator, Muge Dereli, PhD Candidate in Physiotherapy and Rehabilitation, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKCU-IRB-0260; IRB# 0260 (Other: İzmir Katip Çelebi University Health Research Ethics Committee)
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary dysmenorrhea; Menstrual pain; Exercise; Motor imagery; Pain education; Cognition
MeSH Terms: conditions — Dysmenorrhea; Motor Activity | interventions — Resistance Training; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Only (Experimental): Participants will complete an 8-week supervised exercise program including lumbopelvic stabilization, stretching, and endurance training, delivered twice per week.
  Interventions: Behavioral: Exercise Program
- Exercise + Motor Imagery (Experimental): Participants will complete the same 8-week supervised exercise program. In addition, they will practice kinesthetic motor imagery of the exercises before performing them.
  Interventions: Behavioral: Exercise Program; Behavioral: Exercise plus Motor Imagery Training
- Exercise + Pain Neuroscience Education (Experimental): Participants will complete the same 8-week supervised exercise program. In addition, they will receive weekly face-to-face pain neuroscience education sessions supported by home assignments.
  Interventions: Behavioral: Exercise Program; Behavioral: Exercise plus Pain Neuroscience Education

INTERVENTIONS:
Behavioral: Exercise Program — Participants will complete an 8-week supervised exercise program, delivered twice per week. The program includes lumbopelvic stabilization, stretching, and endurance training exercises designed to reduce menstrual pain and improve physical function.
Behavioral: Exercise plus Motor Imagery Training — Participants will complete the same 8-week supervised exercise program as the Exercise Only group. In addition, they will practice kinesthetic motor imagery of the prescribed movements prior to performing them, aiming to enhance motor control and pain modulation.
  Arms: Exercise + Motor Imagery
Behavioral: Exercise plus Pain Neuroscience Education — Participants will complete the same 8-week supervised exercise program as the Exercise Only group. In addition, they will receive weekly face-to-face pain neuroscience education sessions focused on pain neurophysiology, supported with home assignments to reinforce learning.
  Arms: Exercise + Pain Neuroscience Education

SUMMARY:
The goal of this clinical trial is to find out whether exercise, motor imagery training, and pain neuroscience education can help reduce menstrual pain and improve well-being in young women with primary dysmenorrhea. The study will also look at how these approaches affect menstrual symptoms, movement control, and cognitive flexibility.

The main questions it aims to answer are:

* Does adding motor imagery or pain neuroscience education to an exercise program reduce pain and menstrual symptoms more than exercise alone?
* Do these approaches improve movement control, thinking flexibility, and knowledge about pain?

Researchers will compare three groups:

* Exercise only
* Exercise plus motor imagery training
* Exercise plus pain neuroscience education

Participants will:

* Attend supervised exercise sessions twice a week for 8 weeks
* Practice either motor imagery or receive short pain neuroscience education, depending on their group
* Complete questionnaires and tests before and after the program, during the first three days of menstruation

DETAILED DESCRIPTION:
Primary dysmenorrhea is a common gynecological condition characterized by menstrual pain without underlying pathology. It negatively impacts quality of life and may affect cognitive functions such as attention and flexibility. Non-pharmacological interventions such as exercise, motor imagery, and pain neuroscience education are promising approaches for pain management without side effects. However, evidence on their effectiveness in primary dysmenorrhea is limited.

This randomized controlled trial is designed to compare the effects of three different interventions in young women with primary dysmenorrhea:

* Exercise only (control group)
* Exercise plus Motor Imagery Training
* Exercise plus Pain Neuroscience Education (PNE)

Eligible participants will be women aged 18-25 years who meet the diagnostic criteria for primary dysmenorrhea based on gynecological examination and ultrasound findings. Participants will be randomly assigned into one of the three groups. All groups will undergo an 8-week supervised exercise program (two sessions per week) focusing on lumbopelvic stabilization, flexibility, and endurance training. In addition:

* The Motor Imagery group will practice kinesthetic visualization of the exercises prior to performing them.
* The PNE group will receive weekly face-to-face education sessions on pain mechanisms, supported with home assignments.

Primary outcome measures are:

* Pain intensity (Numeric Pain Rating Scale)
* Pressure pain threshold (Baseline dolorimeter)
* Menstrual symptoms (Menstrual Symptom Questionnaire).

Secondary outcome measures are:

* Lumbopelvic motor control (Physiosupplies Core Stabilizer Unit)
* Movement Imagery Questionnaire
* Central Sensitization Inventory
* Cognitive flexibility (Stroop Test)
* Pain Catastrophizing Scale
* Pain Resilience Scale
* Modified Pain Neurophysiology Questionnaire.

Assessments will be conducted at baseline and after the 8-week intervention, within the first three days of menstruation. Additional follow-up data will be collected through online forms one month after the intervention to evaluate persistence of effects.

The estimated sample size of 51 was calculated considering a 10% attrition rate. Statistical analyses will be performed using SPSS software. Depending on data distribution, repeated measures ANOVA or non-parametric equivalents will be used to compare changes over time and between groups.

This study is expected to provide new evidence regarding the effectiveness of combining exercise with motor imagery or pain neuroscience education for the management of pain, menstrual symptoms, and cognitive flexibility in women with primary dysmenorrhea. The findings may contribute to the development of safe and effective non-pharmacological strategies in women's health and pain management.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-25 years
* Gynecological examination and ultrasound confirming absence of pelvic pathology
* History of primary dysmenorrhea for at least 6 months, with pain intensity ≥4 on the Numeric Rating Scale (0-10) during the first 3 days of menstruation
* Regular menstrual cycles (21-35 days)
* Nulliparous (no history of pregnancy or childbirth)
* No systemic, metabolic, rheumatologic, or lumbar pathology
* Willingness to participate in the 8-week intervention program and attend follow-up assessments

Exclusion Criteria:

* Diagnosis of secondary dysmenorrhea (e.g., endometriosis, pelvic inflammatory disease, uterine fibroids, ovarian cysts)
* Current pregnancy or planning to become pregnant during the study period
* History of pelvic or abdominal surgery
* History of sexually transmitted diseases
* Current use of antidepressants, anxiolytics, or hormonal therapy (e.g., oral contraceptives, intrauterine device)
* Known neurological, psychiatric, or systemic musculoskeletal disorders
* Cognitive impairment or attention deficit that may interfere with participation
* Participation in regular exercise in the last 6 months
* Use of alternative therapies for dysmenorrhea (e.g., acupuncture, massage)

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only individuals who self-identify as female and have biological capacity for menstruation (i.e., women of reproductive age with regular menstrual cycles) are eligible to participate.
Enrollment: 51 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline, after 8 weeks of intervention, and 1 month post-intervention follow-up
  Pain intensity will be assessed using an 11-point Numeric Rating Scale (0 = no pain, 10 = worst imaginable pain). Participants will be asked to report their average menstrual pain during the first three days of menstruation.
Pressure Pain Threshold (PPT) | Baseline and after 8 weeks of intervention (first three days of menstruation)
  Pressure pain threshold will be measured using a digital algometer (Baseline dolorimeter) applied to the abdominal region and standardized body sites. The minimum pressure (kg/cm²) at which pain is first perceived will be recorded.
Menstrual Symptom Severity | Baseline, after 8 weeks of intervention, and 1 month post-intervention follow-up
  Menstrual symptoms (e.g., cramps, headache, back pain, fatigue, mood changes) will be evaluated using the Menstrual Symptom Questionnaire (MSQ). Total and subscale scores will be calculated.

SECONDARY OUTCOMES:
Lumbopelvic Motor Control | Baseline and after 8 weeks of intervention
  Lumbopelvic motor control will be assessed using the Physioupplies Core Stabilizer Unit, which measures pressure changes during standardized stabilization tasks.
Movement Imagery Ability | Baseline
  Participants' ability to generate and control movement imagery will be assessed using the Movement Imagery Questionnaire. Higher scores indicate better imagery ability.
Central Sensitization | Baseline, after 8 weeks of intervention, and 1 month post-intervention follow-up
  Central sensitization symptoms will be evaluated using the Central Sensitization Inventory (CSI). The total score reflects symptom severity.
Cognitive Flexibility | Baseline and after 8 weeks of intervention
  Cognitive flexibility and inhibitory control will be assessed using the EncephalApp Stroop application. Participants will complete the "off" and "on" runs. Primary variables will be total completion time (seconds) and error count; lower times and fewer errors indicate better performance.
Pain Catastrophizing | Baseline, after 8 weeks of intervention, and 1 month post-intervention follow-up
  Catastrophic thinking related to pain will be assessed with the Pain Catastrophizing Scale, which includes rumination, magnification, and helplessness subscales.
Pain Resilience | Baseline, after 8 weeks of intervention, and 1 month post-intervention follow-up
  Resilience in response to pain will be measured using the Pain Resilience Scale. Higher scores indicate better psychological resilience.
Pain Neurophysiology Knowledge | Baseline (all groups); post-intervention and 1-month follow-up (PNE group only)
  Participants' knowledge of pain mechanisms will be evaluated using the Revised Neurophysiology of Pain Questionnaire (NPQ). Higher scores indicate greater understanding of pain biology. The questionnaire will be administered to all participants at baseline (before the start of the intervention). In addition, it will be repeated only in the Pain Neuroscience Education (PNE) group immediately after the 8-week intervention and 1 month later to evaluate changes in knowledge.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (pain intensity scores, pressure pain threshold values, questionnaire results, and demographic data) will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 6 months after study completion and will remain available for 5 years.
Access Criteria: Researchers who provide a methodologically sound proposal will be able to access the data for academic purposes. Data will be shared via email request to the principal investigator, subject to approval by the study team.

REFERENCES:
- [Background] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Background] Evans S, Dowding C, Olive L, Payne LA, Druitt M, Seidman LC, Skvarc D, Mikocka-Walus A. Pain catastrophizing, but not mental health or social support, is associated with menstrual pain severity in women with dysmenorrhea: A cross-sectional survey. Psychol Health Med. 2022 Jul;27(6):1410-1420. doi: 10.1080/13548506.2021.1948581. Epub 2021 Jun 30. PMID 34190659
- [Background] Cuenca-Martinez F, Nieves-Gomez A, Millan-Isasi N, Fuentes-Aparicio L, Sempere-Rubio N. Effects of motor imagery and action observation on pelvic floor and related structures in healthy women: A randomized controlled trial. Hum Mov Sci. 2025 Feb;99:103313. doi: 10.1016/j.humov.2024.103313. Epub 2024 Dec 2. PMID 39626586
- [Background] Kluska J, Malinowska E, Kowalski J. A pilot longitudinal study of decrease in cognitive functions during the most painful day of the period among women with primary dysmenorrhea. Arch Gynecol Obstet. 2025 Feb;311(2):341-346. doi: 10.1007/s00404-024-07617-9. Epub 2024 Jul 4. PMID 38963585
- [Background] Carroquino-Garcia P, Jimenez-Rejano JJ, Medrano-Sanchez E, de la Casa-Almeida M, Diaz-Mohedo E, Suarez-Serrano C. Therapeutic Exercise in the Treatment of Primary Dysmenorrhea: A Systematic Review and Meta-Analysis. Phys Ther. 2019 Oct 28;99(10):1371-1380. doi: 10.1093/ptj/pzz101. PMID 31665789